CLINICAL TRIAL: NCT01861522
Title: A Confirmatory Study of TAU-284 in Pediatric Patients With Perennial Allergic Rhinitis (A Randomized, Double-blind, Placebo-controlled Study)
Brief Title: The Confirmatory Study of TAU-284 in Pediatric Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAU-284-20
Record Dates: First submitted 2013-05-19; First posted 2013-05-23 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Perennial Allergic Rhinitis
Keywords: TAU-284; Bepotastine besilate; Histamine H1 receptor antagonists; children
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — bepotastine besilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU-284 (Experimental): Two TAU-284 5mg tablets will be taken orally twice a day, once after breakfast and once after dinner (or before bed).
  Interventions: Drug: Bepotastine besilate
- Placebo (Placebo Comparator): Two placebo tablets will be taken orally twice a day, once after breakfast and once after dinner (or before bed).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bepotastine besilate — Two TAU-284 5mg tablets will be taken orally twice a day
  Other Names: TALION 5mg tablets
  Arms: TAU-284
Drug: Placebo — Two Placebo tablets will be taken orally twice a day
  Arms: Placebo

SUMMARY:
The objectives of this study are: to confirm the superiority of TAU-284 over placebo after two weeks of administration to pediatric patients with perennial allergic rhinitis and to investigate safety of TAU-284.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 2-arm parallel-group comparative study to confirm the superiority of TAU-284 over placebo after two weeks of administration of TAU-284 (20 mg/day) or placebo to pediatric patients with perennial allergic rhinitis, with "the change from baseline in total nasal symptom score (total score for the three major nasal symptoms [sneezing, rhinorrhea, and nasal congestion])" as the primary endpoint; and to investigate safety of TAU-284.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 7 and 15 years
* Patients who have received a diagnosis of perennial allergic rhinitis according to the diagnostic criteria
* Patients with a mean rhinorrhea score and a mean sneezing score of at least 2 on the basis of symptoms recorded in the nasal allergy diary during the observation period etc.

Exclusion Criteria:

* Patients with vasomotor rhinitis or eosinophilic rhinitis
* Patients who have concurrent nasal disease that may affect the efficacy of TAU-284
* Patients with a history of any of the nasal surgical procedures
* Patients who have a positive result for pollen antigens which are dispersed during the study period
* Patients who have a positive result for dog dander or cat dander antigen and have a chance to touch dogs or cats.
* Patients with current or previous history of drug allergy
* Patients who concurrently have renal function abnormalities that may cause safety problems etc.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 473 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KIMIHIRO OKUBO, Study Director — Nippon Medical School
Locations (2):
- Japan (2):
  - Reserch site, Fukuoka
  - Reserch site, Toyama

REFERENCES:
- [Result] Okubo K, Ichimura M, Koyama T, Susuta Y, Izaki H. Double-blind placebo-controlled study of bepotastine besilate in pediatric patients with perennial allergic rhinitis. Expert Opin Pharmacother. 2015;16(16):2395-408. doi: 10.1517/14656566.2015.1085511. Epub 2015 Sep 12. PMID 26364765

RESULTS

PARTICIPANT FLOW:
Groups:
- TAU-284: TAU-284 10mg twice daily for 2 weeks
- Placebo: TAU-284 placebo twice daily for 2 weeks
Period: Overall Study
Arm/Group | TAU-284 | Placebo
Started | 240 | 232 (One subject who did not receive any study drug was excluded from the FAS and the Safety Analysis Set)
Completed | 237 | 232
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAU-284 | Placebo | Total
Number analyzed (Participants) | 240 | 232 | 472
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (2.4) | 10.4 (2.4) | 10.4 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 92 | 200
  Male | 132 | 140 | 272

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score for the Three Major Nasal Symptoms [Sneezing, Rhinorrhea, and Nasal Congestion]
Description: Total score for the three major nasal symptoms (sneezing, rhinorrhea, and nasal congestion) were rated on 5-point scale ranging from 0 (no symptoms) to 4 (very severe).
Time Frame: Baseline and Week 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TAU-284 | Placebo
Number analyzed (Participants) | 240 | 232
units on a scale | -1.579 (0.090) | -1.110 (0.092)

2. Secondary Outcome: Change From Baseline in Total Score for the Three Major Nasal Symptoms [Sneezing, Rhinorrhea, and Nasal Congestion]
Time Frame: baseline, Week1 and Week 2
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Individual Nasal Symptom Scores (Sneezing, Rhinorrhea, Nasal Congestion, and Impairment in Daily Activities)
Time Frame: baseline, Week1 and Week 2
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Individual Scores for Local Nasal Findings (Rhinoscopic Findings)
Time Frame: baseline, Week1 and Week 2
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Severity Score for Symptoms of Allergic Rhinitis
Time Frame: Randomization, Week1 and Week 2
Reporting Status: Not Posted

6. Secondary Outcome: Adverse Events and Adverse Drug Reactions
Time Frame: Week 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | TAU-284 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/232
Other Adverse Events (participants affected / at risk) | 17/240 | 15/232
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAU-284 (N=240) | Placebo (N=232)
Pharyngitis (Infections and infestations) | 10 | 6
Nasopharyngitis (Infections and infestations) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other